CLINICAL TRIAL: NCT01974531
Title: Psychological Distress & Stress in Parents With Preterm infants-a Prospective Study on Risk and Protective Psychobiological Aspects
Brief Title: Psychological Distress & Stress in Parents With Preterm infants-a Prospective Study
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Goethe University (Other)
Responsible Party: Principal Investigator, Dr. Silvia Oddo, PhD, Johann Wolfgang Goethe University Hospital
Other Study IDs: Louwen/Oddo-Preterm birth
Record Dates: First submitted 2013-10-28; First posted 2013-11-01 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Preterm Birth; Pregnancy; Stress; Psychological Distress
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm birth/ Timely birth
- Women/men

SUMMARY:
The purpose of the present prospective study is the analysis of risk and protective factors of perinatal stress and psychological distress of parents with or without a preterm child. Stress is measured biologically by Cortisol levels and psychologically by a questionnaire. Different outcomes of psychological distress (e.g. anxiety, depression, posttraumatic stress disorder, burnout) are measured by various questionnaires. We analyze the influence of different aspects as personality traits, social support, partnership.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women and their partners from the 24th week of gestation on
* 18 years of age

Exclusion Criteria:

* psychiatric, mainly psychotic diseases
* drug abuse
* severe neurological disorders
* stillbirth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women either with risk of with no risk of preterm birth from the obstetric ward or from the antenatal class of the obstetric department and their partners
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
stress | two years

CONTACTS AND LOCATIONS:
Overall Officials: Frank Louwen, Prof., Study Director — University Hospital Frankfurt-Dept. Obstetrics and Perinatal Medicine
Locations (1):
- University Hospital Frankfurt-Dept.Obstetrics and Perinatal Medicine, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Sommerlad S, Schermelleh-Engel K, La Rosa VL, Louwen F, Oddo-Sommerfeld S. Trait anxiety and unplanned delivery mode enhance the risk for childbirth-related post-traumatic stress disorder symptoms in women with and without risk of preterm birth: A multi sample path analysis. PLoS One. 2021 Aug 31;16(8):e0256681. doi: 10.1371/journal.pone.0256681. eCollection 2021. PMID 34464408